CLINICAL TRIAL: NCT05207020
Title: Study Allowing the Collection of Clinical and Biological Data Necessary for Development and Validation of the Blood Glucose Measurement Device by Air Analysis Expired Developed by the Company BOYDSense
Brief Title: Development and Validation of the Blood Glucose Measurement Device by Air Analysis Expired
Acronym: BOYDSENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/21/0305
Record Dates: First submitted 2021-11-30; First posted 2022-01-26 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; self monitoring of blood glucose,; breath glucose monitoring system
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Single group with a device
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sugar levels estimated by analysis of exhaled air (Experimental)
  Interventions: Device: Glycemia estimated by exhaled air analyzer; Behavioral: Questionnaire; Biological: Veinous glycemia; Biological: Capillary glycemia; Biological: constitution biological collection; Biological: Blood sample; Other: Test meal

INTERVENTIONS:
Device: Glycemia estimated by exhaled air analyzer — Measurement of volatile compounds in the air exhaled by the volunteer on 3 different MIBs (3 breaths in total) at 7 times: T0, 30min, 1H, 1H30, 2H, 2H30, 3H after test meal
Behavioral: Questionnaire — The questionnaire focuses on the methods and feelings of the blood glucose self-monitoring that he is currently carrying out, a first feedback on user experience on the operation of the prototype and the collection of his expectations for a future commercial device
Biological: Veinous glycemia — Measurement of the veinous glycemia at 7 times: T0, 30min, 1H, 1H30, 2H, 2H30, 3H after test meal
Biological: Capillary glycemia — 7-step capillary glycemia measurement: T0, 30min, 1H, 1H30, 2H, 2H30, 3H after test meal
Biological: constitution biological collection — Sampling for storage of serum at 7 times: T0, 30min, 1H, 1H30, 2H, 2H30, 3H after test meal
Biological: Blood sample — Single blood sample before mealtimes for HbA1C molecular analysis
Other: Test meal — taking a test meal before the various blood sugar measurements

SUMMARY:
This clinical study aims to finalize the algorithm and assess the performance of the BOYDSense® breath glucose monitoring system prototype in patients living with type 2 diabetes.

DETAILED DESCRIPTION:
Self-monitoring of blood glucose (SMBG) is prescribed to patients living with diabetes according to their type of diabetes, their clinical profile and their personalized needs such as therapeutic adjustments, detection of an asymptomatic hyperglycaemic drift, prevention of hypoglycaemia, or adaptation of the therapeutic strategy to the evolution of the pathology. Most of the people living with type2 diabetes mellitus (T2DM) use an invasive finger prick SMBG glucometer. A pilot study conducted by the BOYDSense mother company Alpha-MOS showed that the analysis of volatile organic compounds (VOC) in exhaled air could reliably predict blood glucose. The development of a breath glucose-monitoring device, by its non-invasive nature, should be an alternative to existing systems by making it possible to avoid capillary samples. Investigators could expect a better quality of life and a better compliance with SMBG in the majority of patients with T2DM. The objectives of our study are to improve the BOYDSense®glucose algorithm based on the VOC analysis of exhaled air; then to assess the performance of the BOYDSense® prototype with the finalized algorithm.

This study aims to gather, in patients with T2DM, successive blood and capillary reference glucose values during a meal test, and to compare them to glucose levels estimated by the BOYDSense® prototype.

All the enrolled patients will undergo a 3 hours standardized meal test with seven glucose measurement endpoints at T0, 30 min, 1hour 1H30, 2H, 2H30 and 3H post meal. Blood glucose will be measured with three different techniques: venous blood glucose measured with a COBAS 8000 automatic analyzer, SMBG measured with a commercial glucometer and blood glucose value estimated from exhaled air using the BOYDSense® prototype.

The study duration will be 4H for each enrolled patient. After the meal test being completed, the end of study procedure includes a 30 min observational period dedicated to the completion of the patients'questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed for at least 3 months.
* Acceptance of constraints related to participation in the study.
* Acceptance to participate in the constitution of a plasma library.
* Ability to sign informed consent.
* Affiliation to a social security scheme.

Exclusion Criteria:

* Ongoing prandial insulin therapy
* Treated bacterial or viral respiratory infection in the 2 weeks preceding the meal test.
* Surgical intervention under general anesthesia in the last 12 weeks.
* Asthmatic subjects with bronchospasm or under chronic inhaled therapy.
* Ongoing COVID-19 (PCR +) or contact case in the isolation period.
* Pregnancy or breast-feeding.
* Participation in another clinical study or exclusion period from another research protocol.
* Patient under guardianship, curatorship or legal protection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Collect glucose values | 1 day
  Collect successive fasting blood glucose values in patients with type 2 diabetes
Collect glucose values | 1day
  Collect successive blood glucose values after taking a test meal, in patients with type 2 diabetes
Collect glucose values (fasting) | 1 day
  Measurement of blood glucose by the exhaled air analyzer from volatile compounds in exhaled air (fasting)
Collect glucose values (after a test meal) | 1 day
  Measurement of blood glucose by the exhaled air analyzer from volatile compounds in exhaled air (after taking a test meal))

CONTACTS AND LOCATIONS:
Overall Officials: Pierre GOURDY, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service de Diabétologie, maladies métaboliques et nutrition, CHU Toulouse, 1 avenue Jean Pouilhes, TSA 50032, Toulouse, France

IPD SHARING:
Plan to Share IPD: No